CLINICAL TRIAL: NCT00407563
Title: A Phase 2 Study of Bevacizumab With Abraxane in Patients With Recurrent, Platinum-Resistant Primary Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Bevacizumab With Abraxane in Patients With Recurrent Ovarian/ Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Genentech, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACORN ALSSOPR0501
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-03

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Bevacizumab; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be given via IV infusion at 10mg/kg given on days 1 and 15 of a 28-day cycle.
  Other Names: Avastin
Drug: Abraxane — Abraxane will be given via IV infusion at 100mg/m²over 30 minutes on days 1, 8, and 15 of a 28-day cycle.
  Other Names: albumin-bound paclitaxel

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability of the combination of bevacizumab and Abraxane in the treatment of women with epithelial ovarian cancer or peritoneal cancer. The study will also evaluate how the patient's quality of life is during their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease by CT or MRI.
* At least 1 "target lesion" to be used to assess response as defined by GOG RECIST criteria.
* ECOG performance status of 0 or 1.
* Patient provides voluntary written informed consent.
* At least 18 years of age.
* Negative serum pregnancy test.
* Recovered from any recent surgery for at least 30 days and is free of active infection.
* Received the following prior therapy at time of enrollment:
* Must have had 1 prior platinum-based chemotherapeutic regimen containing carboplatin, cisplatin or organoplatinum. Initial therapy may have included high-dose therapy, consolidation, or extended therapy. Patient should be defined as recurrent or progression of disease within 6 months of last platinum chemotherapy.
* May have had 1 additional cytotoxic or non-cytotoxic chemotherapy regimen.
* Must have adequate hematologic and hepatic function.

Exclusion Criteria:

* Previously received bevacizumab.
* History of other invasive malignancy with the exception of nonmelanoma skin cancer.
* ECOG performance status of 2, 3, or 4.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study. Patient must be bevacizumab naïve.
* Blood pressure of >150/100 mm Hg on antihypertensive medications.
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* Diagnosed with unstable angina per NYHA or Grade 2 or greater congestive heart failure.
* History of myocardial infarction within 6 months of enrollment.
* History of stroke or transient ischemic attack within 6 months prior to study enrollment.
* Clinically significant vascular disease (e.g., aortic aneurysm, aortic dissection)or symptomatic peripheral vascular disease.
* Bleeding diathesis or coagulopathy.
* Presence of CNS or brain metastases.
* Pre-existing peripheral neuropathy of Grade ≥ 2.
* A major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study.
* A partial or complete small or large bowel obstruction demonstrated radiologically within 3 months prior to study enrollment.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment.
* Positive pregnancy test or is lactating.
* History of abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months prior to study enrollment.
* Serious, non-healing wound, ulcer, or bone fracture.
* Serious intercurrent medical or psychiatric illness, including serious active infection.
* Inability to comply with study and/or follow-up procedures.
* Life expectancy of less than 12 weeks.
* Proteinuria at screening as demonstrated by either:
* Urine protein:creatinine (UPC) ratio ≥ 1.0 at screening OR
* Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Schwartzberg, MD, FACP, Principal Investigator — The West Clinic
Locations (11):
- United States (11):
  - Little Rock Hematology Oncology, Little Rock, Arkansas
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Southeastern Gynecologic Oncology, LLC, Atlanta, Georgia
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Hematology-Oncology Centers of the Northern Rockies, Billings, Montana
  - Mid-Ohio Oncology/Hematology, Columbus, Ohio
  - Pennsylvania Oncology Hematology Assoc., Philadelphia, Pennsylvania
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Cancer Specialists of Tidewater, Ltd, Chesapeake, Virginia

REFERENCES:
- [Derived] Tillmanns TD, Lowe MP, Walker MS, Stepanski EJ, Schwartzberg LS. Phase II clinical trial of bevacizumab with albumin-bound paclitaxel in patients with recurrent, platinum-resistant primary epithelial ovarian or primary peritoneal carcinoma. Gynecol Oncol. 2013 Feb;128(2):221-8. doi: 10.1016/j.ygyno.2012.08.039. Epub 2012 Sep 5. PMID 22960352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 community oncology research sites across the US within the ACORN network participated in this study. Enrollment started in January 2007 and was completed in December 2008.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent screening procedures to verify eligibility.
Groups:
- Bevacizumab and Abraxane: All subjects received treatment with bevacizumab and Abraxane. Bevacizumab will be given via IV infusion at 10 mg/kg given on days 1 and 15 of a 28-day cycle. Abraxane will be given via IV infusion at 100 mg/m^2 over 30 minutes on days 1, 8, and 15 of a 28-day cycle.
Period: Overall Study
Arm/Group | Bevacizumab and Abraxane
Started | 48
Completed | 47 (One patient remains on study treatment.)
Not Completed | 1
Not completed — Patient continues on treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Abraxane
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-Free Rate
Description: Progression-free rate is defined as the percentage of participants with no progression event at 6 months after starting study treatment. An event for this endpoint was defined as a progression-free survival event occurring earlier than six months, or discontinuation of treatment earlier than six months for any other reason. Progression is defined per RECIST criteria v1.0 as a measurable increase in the smallest diameter of any target lesion, progression of existing non-target lesions, or the appearance of 1 or more new lesions.
Time Frame: 6 months after initiation of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bevacizumab and Abraxane
Number analyzed (Participants) | 48
percentage of patients | 62.5 [47.8 to 77.2]

2. Secondary Outcome: Best Overall Response
Description: Radiologic imaging was scheduled to be performed at baseline, after every third treatment cycle, and at the end of treatment or time of progression unless it was done in the previous four weeks. Response was evaluated using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; overall response (OR) = CR+PR.
Time Frame: Radiologic imaging was repeated after every 3 cycles (about every 12 weeks) during study treatment, up to 31 months.
Measure: Number; unit: Participants
Arm/Group | Bevacizumab and Abraxane
Number analyzed (Participants) | 48
Participants
  Complete response | 4
  Partial response | 20
  Stable disease | 14
  Progressive disease | 8
  Not evaluable | 2

3. Secondary Outcome: Overall Survival
Time Frame: Overall survival is defined as the time from treatment start until death from any cause, assessed up to 40 months.
Population: Participants who had not experienced death during or after stopping treatment were censored in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Abraxane
Number analyzed (Participants) | 48
Months | 17.15 [13.57 to 23.82]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Disease progression was determined through radiology imaging measurements and by clinical or symptomatic progression during or after treatment. Progression is defined per RECIST criteria v1.0 as a measurable increase in the smallest diameter of any target lesion, progression of existing non-target lesions, or the appearance of 1 or more new lesions.
Time Frame: PFS was measured from day 1 of treatment until time of progression (assessed every 12 weeks) or death, whichever came first, assessed up to 30 months.
Population: Participants who had not experienced either disease progression or death during or after stopping treatment were censored in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Abraxane
Number analyzed (Participants) | 48
Months | 8.08 [5.78 to 10.15]

5. Secondary Outcome: Best Overall Response at Six Months
Description: The outcome measure assessed the percentage of participants who had achieved either a Partial or Complete Response over 6 months of treatment. Radiologic imaging was scheduled to be performed at baseline, after every third treatment cycle, and at the end of treatment or time of progression unless it was done in the previous four weeks. Response was evaluated using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; overall response (OR) = CR+PR.
Time Frame: Assessed over 6 months of study treatment
Population: The 2 tailed, 95% confidence interval of the estimated response rate was calculated using the normal approximation to the binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bevacizumab and Abraxane
Number analyzed (Participants) | 48
percentage of patients | 50 [34.8 to 65.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning on day 1 of study treatment until one month after the end of study treatment, up to 32 months.
Description: Systematic Assessment - subjects were assessed for adverse events weekly by either the research coordinator, treating physician, or other appropriate sub-investigator.
Arm/Group | Bevacizumab and Abraxane
Serious Adverse Events (participants affected / at risk) | 13/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and Abraxane (N=48)
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 1
Hernia obstructive (General disorders) | 1
Pain (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Overdoses (Injury, poisoning and procedural complications) | 1
Body temperature increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and Abraxane (N=48)
Anemia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Erythema of eyelid (Eye disorders) | 2
Eye hemorrhage (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 4
Photopsia (Eye disorders) | 2
Vision blurred (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 5
Feces hard (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 18
Oral pain (Gastrointestinal disorders) | 1
Paresthesia oral (Gastrointestinal disorders) | 1
Peritoneal and retroperitoneal disorders (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1
Reflux gastritis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Sore mouth (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 11
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 14
Asthenia (General disorders) | 1
Catheter site inflammation (General disorders) | 1
Chest pain (General disorders) | 4
Chills (General disorders) | 4
Fatigue (General disorders) | 37
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site reaction (General disorders) | 1
Local swelling (General disorders) | 2
Localized edema (General disorders) | 2
Malaise (General disorders) | 1
Nodule (General disorders) | 1
Edema peripheral (General disorders) | 3
Pain (General disorders) | 5
Pyrexia (General disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Multiple allergies (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Localized infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 2
Pharyngitis streptococcal (Infections and infestations) | 1
Postpoperative wound infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sepsis syndrome (Infections and infestations) | 1
Sialoadenitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 7
Streptococcal infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 11
Vaginal infection (Infections and infestations) | 2
Vaginitis bacterial (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 2
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 3
Skin laceration (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Blood pressure increased (Investigations) | 2
Blood thyroid stimulating hormone increased (Investigations) | 1
Body temperature increased (Investigations) | 4
C-reactive protein increased (Investigations) | 1
CD4 lymphocytes increased (Investigations) | 1
Forced expiratory volume (Investigations) | 1
Hematocrit decreased (Investigations) | 1
Hemoglobin decreased (Investigations) | 2
Monoctye count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Parasite stool test positive (Investigations) | 1
Platelet count decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Weight loss poor (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Foot fracture (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 7
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 12
Hypoesthesia (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 3
Nerve compression (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 15
Paresthesia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 2
Disturbance in attention (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 9
Mood altered (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 6
Hematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 6
Urethral pain (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Edema genital (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 3
Vulvovaginal pruritis (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder, NOS (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 15
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 4
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Skin discoloration (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Umbilical hemorrhage (Skin and subcutaneous tissue disorders) | 1
Ileostomy (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 10
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publication must be submitted to Funder at least 60 days prior to the submission for publication. If Funder requests in writing, the proposed publication may be held for an additional 90 days.